CLINICAL TRIAL: NCT04946318
Title: A 24-week, Multicenter, Randomized, Double-blind, Parallel-arm, Placebo-controlled Extension Study to Assess the Safety of CSJ117, When Added to Existing Standard of Care Asthma Therapy in Patients ≥18 Years of Age
Brief Title: Study of Safety of CSJ117 in Participants With Moderate to Severe Uncontrolled Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCSJ117A12201E1; 2020-002341-42 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Asthma
Keywords: CSJ, GINA 2019, Safety
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 24-week Placebo (Placebo Comparator): Participants who will enter the extension study after the last treatment visit (week 12) of the core study and will be treated with Placebo inhaled once daily for 24 weeks
  Interventions: Drug: CSJ117; Drug: Placebo
- 12-week wash out + 12-week Placebo (Placebo Comparator): Participants who will enter the extension study after the last treatment visit (week 12) of the core study and will be treated with Placebo inhaled once daily for 12 weeks "washout period" and Placebo inhaled once daily for 12 weeks
  Interventions: Drug: CSJ117
- 12-week Placebo (Placebo Comparator): Participants who will enter the extension study after the last follow-up visit (week 24) of the core study will be treated with Placebo inhaled once daily for 12 weeks
  Interventions: Drug: CSJ117
- 24-week CSJ117 (Experimental): Participants who will enter the extension study after the last treatment visit (week 12) of the core study and will be treated once daily for 24 weeks with the same dose of CSJ117 they received in the core study. CSJ117 (0.5 mg, 1 mg, 2 mg, 4 mg and 8 mg) inhaled once daily for 24 weeks.
  Interventions: Drug: CSJ117
- 12-week wash out + 12-week CSJ117 (Experimental): Participants who will enter the extension study after the last treatment visit (week 12) of the core study and will be treated with Placebo inhaled once daily for 12 weeks "washout period" and then they will be treated once daily for 12 weeks with the same dose of CSJ117 they received in the core study. CSJ117 (0.5 mg, 1 mg, 2 mg, 4 mg and 8 mg) inhaled once daily for 12 weeks.
  Interventions: Drug: CSJ117
- 12-week CSJ117 (Experimental): Participants who will enter the extension study after the last follow-up visit (week 24) of the core study will be treated with once daily for 12 weeks with the same dose of CSJ117 they received in the core study. CSJ117 (0.5 mg, 1 mg, 2 mg, 4 mg and 8 mg) inhaled once daily for 24 weeks.
  Interventions: Drug: CSJ117

INTERVENTIONS:
Drug: CSJ117 — CSJ117 (0.5 mg, 1mg, 2mg, 4 mg and 8 mg) capsules for inhalation once daily delivered via Concept1 inhalation device for 12 or 24 weeks.
Drug: Placebo — Placebo inhaled once daily for 12 or 24 weeks. Delivered via Concept1 device.
  Arms: 24-week Placebo

SUMMARY:
The purpose of this study is to provide safety and tolerability, pharmacokinetics and immunogenicity data for multiple CSJ117 doses inhaled once daily compared with placebo, in adult asthma participants treated with medium or high dose ICS plus LABA alone or with additional asthma controllers (additional controllers allowed: LTRA, LAMA, Theophylline and its derivatives), who have completed the prior phase llb study CCSJ117A12201C (NCT04410523).

DETAILED DESCRIPTION:
This is a 12/24-week Phase llb, multicenter, multi-national, double-blind, randomized, parallel-arm, placebo-controlled extension study to evaluate the safety and tolerability, pharmacokinetics and immunogenicity of 5 dose levels of CSJ117 in adult asthma participants treated with medium or high dose ICS plus LABA alone or with additional asthma controllers (allowed: LTRA, LAMA, theophylline or its derivatives), who have completed the prior core phase llb study CCSJ117A12201C (NCT04410523). The study will include the following three parts:

A Screening period of up to 3 days to assess eligibility.

A Treatment period of 12 or 24 weeks. There are two scenarios on when a participant can enroll into the extension study depending on when the study site is activated for the extension study CCSJ117A12201E1:

* A 24 week treatment period: Participants on each of the five treatment arms (CSJ117 0.5 to 8 mg) or placebo of the core study CCSJ117A12201C, who will enter the extension study after the last Treatment period visit (week 12) of the core study, will be randomized in a 1:1 ratio to continue on their previously assigned CSJ117 dose or placebo from CCSJ117A12201C for 24 weeks, or to first go through a 12-week "washout period" receiving placebo (for the blinding purpose) and then restart on their previously assigned CSJ117 dose or placebo from CCSJ117A12201C for 12 weeks.
* A 12 week treatment period: Participants on each of the five treatment arms (CSJ117 0.5 to 8 mg) or placebo of the core study CCSJ117A12201C, who will enter the extension study after the last Follow-up visit (week 24) of the core study, will restart on their previously assigned CSJ117 dose or placebo from CCSJ117A12201C for 12 weeks.

A Follow-up period of 12 weeks, study drug free, following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have been treated with a fixed dose combination of fluticasone propionate/salmeterol in one of two doses in stable dose alone or with additional controllers at label approved dosage (allowed only: LTRA, LAMA, Theophylline or its derivatives).
* Participants completing the Treatment period and Follow-up period of study CSJ117A12201C and continuing with study CCSJ117A12201E1 must have completed the Treatment period of CSJ117A12201C (i.e. did not discontinue blinded study treatment prematurely) and Follow-up period of study CSJ117A12201C.

Exclusion Criteria:

* Participants who were enrolled into prior study CSJ117A12201C and developed a significant and/or permanent health condition during the prior study.
* Participants who experienced a serious and drug-related AE in the prior study CSJ117A12201C.
* Participants receiving any prohibited medications.
* Participants with a history or current diagnosis of ECG abnormalities.
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (AEs) and serious adverse events (SAEs) | From start of treatment in the core study and until 30 days after end of treatment in the extension study. Up to 40 weeks.
  Number of treatment emergent AEs, AEs leading to study treatment discontinuation, SAEs and SAEs leading to study treatment discontinuation.
  Treatment emergent AEs and SAEs will be counted from first day of treatment of the core study (CCSJ117A12201C) and until 30 days after last day of treatment in the extension study. For participants who will enter the extension study after the last follow-up visit (week 24) of the core study, AEs (if any) occurring from week 4 to week 12 of the drug free follow-up period will not be counted as treatment emergent AEs.
Number of treatment emergent participant deaths and participant hospitalizations | From start of treatment in the core study and until 30 days after end of treatment in the extension study. Up to 40 weeks.
  Number of treatment emergent participant deaths and participant hospitalizations (any visit to the hospital requiring an overnight stay or an emergency room visit greater than 24 hours).
  Treatment emergent participant deaths and participant hospitalizations will be counted from first day of treatment of the core study (CCSJ117A12201C) and until 30 days after last day of treatment in the extension study. For participants who will enter the extension study after the last follow-up visit (week 24) of the core study, participant deaths and hospitalizations (if any) occurring from week 4 to week 12 of the drug free follow-up period will not be counted as treatment emergent participant deaths and hospitalizations.

SECONDARY OUTCOMES:
Trough plasma concentration (Ctrough) at Steady State | Participants entering directly after completion of study treatment of core study: Weeks 2, 4, 8, 12, 14, 16, 20, 24, 26, 28 and 36; Participants entering directly after completion of the core study Follow-up period: Weeks 2, 4, 8, 12, 14, 16 and 24.
  Ctrough measured during the treatment period and the follow up period.
Terminal Elimination half-life (T1/2) at Steady State | Participants entering directly after completion of study treatment of core study: Weeks 2, 4, 8, 12, 14, 16, 20, 24, 26, 28 and 36; Participants entering directly after completion of the core study Follow-up period: Weeks 2, 4, 8, 12, 14, 16 and 24.
  Terminal Elimination half-life (T1/2) measured during the treatment period and the follow up period.
Change from baseline in Anti-drug immune response | Participants entering directly after completion of study treatment of core study: Weeks 2, 4, 8, 12, 14, 16, 20, 24, 26, 28 and 36; Participants entering directly after completion of the core study Follow-up period: Weeks 2, 4, 8, 12, 14, 16 and 24.
  The change from baseline in Anti-Drug Antibodies (ADA) titers during the treatment period and the follow up period.
Change from baseline in Fractional exhaled Nitric Oxide (FeNO) levels | Participants entering directly after completion of study treatment of core study: Weeks 2, 4, 8, 12, 14, 16, 20, 24, 26, 28 and 36; Participants entering directly after completion of the core study Follow-up period: Weeks 2, 4, 8, 12, 14, 16 and 24.
  The change from baseline (same as in the core study CSJ117A12201C) in the observed values in FeNO (including all scheduled post-baseline visits with FeNO data).
CSJ117 serum concentration | Participants entering directly after completion of study treatment of core study: Weeks 2, 4, 8, 12, 14, 16, 20, 24, 26, 28 and 36; Participants entering directly after completion of the core study Follow-up period: Weeks 2, 4, 8, 12, 14, 16 and 24.
  Measurement of the total CSJ117 serum concentration during the treatment period and the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (9):
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, White Marsh, Maryland
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, McKinney, Texas
- Argentina (6):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ranelagh, Partido de Berazate, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Paraná
- Novartis Investigative Site, Erpent, Belgium
- Bulgaria (2):
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Stara Zagora
- Canada (3):
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Lovosice
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Witten
- Hungary (3):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Komárom
- Japan (10):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Setagaya-Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Toshima City, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
  - Novartis Investigative Site, Osaka
- Latvia (3):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Philippines (2):
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Manila
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
- Russia (2):
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
- Novartis Investigative Site, Levice, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com